CLINICAL TRIAL: NCT02243085
Title: Predictors of de Novo Urge Urinary Incontinence After Photoselective Vaporization of the Prostate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Min Chul Cho, Assistant professor, DongGuk University
Other Study IDs: MCho2
Record Dates: First submitted 2014-09-13; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia; Urgency; Urinary Incontinence
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- photoselective vaporization

SUMMARY:
The aim of this study was to investigate the incidence of de novo urge urinary incontinence after the photoselective vaporization of the prostate for benign prostatic hyperplasia using the validated overactive bladder symptom score, and to determine the predictors of de novo urge urinary incontinence following the photoselective vaporization of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* men in whom 6-months follow-up data were available
* men who did not complain of urge urinary incontinence based on the OABSS (overactive symptom score): OABSS question 4 score of ≤ 1

Exclusion Criteria:

* previous prostate or bladder surgery
* a previous diagnosis of urethral stricture or prostate carcinoma or bladder cancer or neurogenic bladder disease

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who underwent photoselective vaporization of the prostate using 80 watt potassium-titanyl-phosphate (KTP) laser or 120 watt high-power-system (HPS) laser for benign prostatic hyperplasia refractory to medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
de novo urge urinary incontinence at 6 months after surgery | 6 months postoperatively
  de novo urge urinary incontinence: OABSS (overactive bladder symptom score) question 4 of ≥ 2

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Cho, M.D., Ph.D., Principal Investigator — DongGuk University
Locations (1):
- Dongguk University ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea